CLINICAL TRIAL: NCT02231112
Title: Feasibility of Prone Position in Postoperative Whole Breast Radiation Therapy in Korean Breast Cancer Patient
Brief Title: Whole Breast RT on Prone Position in Korean Women
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Doo Ho Choi, Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-06-138-001
Record Dates: First submitted 2014-08-25; First posted 2014-09-04 (Estimated); Last update posted 2014-11-07 (Estimated); Status verified 2014-11

CONDITIONS: Breast Cancer
Keywords: Korean; Left side
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Prone position whole breast RT (Experimental)
  Interventions: Radiation: Whole breast RT on prone position

INTERVENTIONS:
Radiation: Whole breast RT on prone position

SUMMARY:
It is well known fact that postoperative whole breast radiation therapy (RT) in left breast cancer patient can cause cardiac problem according to the exposed dose. In the several studies in other countries, it was repeatedly showed that RT on prone position can reduce cardiac exposed RT dose in left breast cancer. However, the effectiveness of prone position in RT is not studied in the Korean women have relatively small breast. The investigators planned this study to evaluate the real efficacy of prone position in Korean breast cancer treated with RT.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed left breast cancer
* 20 or older age
* less than 70 years old
* after curative resection
* Eastern Cooperative Oncology Group performance status 0 to 1
* Informed consent to this study
* Consent to contraception for 6 months after RT completion

Exclusion Criteria:

* Male breast cancer
* Combined distant metastasis
* Status of pregnant or brest feeding
* Previous RT history of chest or neck area
* Indication of supraclavicular RT
* Not indicated postoperative whole breast RT

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Irradiated cardiac dose | At simulation, expected average of 1 week

SECONDARY OUTCOMES:
Irradiated dose of left anterior descending artery | At simulation, expected average of 1 week
Irradiated lung dose | At simulation, expected average of 1 week
Clinical target volume (volume, homogeneity index, conformity index) | At simulation, expected average of 1 week
Irradiated dose of axillary lymphatic area | At simulation, expected average of 1 week
Skin change after RT | At 3 months after RT completion
Breast shape after RT | At 6 months after RT completion

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea